CLINICAL TRIAL: NCT00147381
Title: Effectiveness and Safety of Campath-1H as an Induction Agent in Combination With Tacrolimus Monotherapy for Prevention of Graft Rejection Compared to Tacrolimus in Combination With MMF and Steroids in Cadaveric Kidney Transplantation
Brief Title: Effectiveness and Safety of Campath in Combination With Tacrolimus Monotherapy to Prevent Kidney Graft Rejection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Dr. Claudia Bösmüller (Other)
Collaborators: Astellas Pharma GmbH (Industry)
Responsible Party: Sponsor-Investigator, Dr. Claudia Bösmüller, Dr. med., Medical University Innsbruck
Organization: Medical University Innsbruck (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TaCam 07_MC; DE-02-RG-121/Margreiter
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Kidney Transplantation
Keywords: Campath-1H; Alemtuzumab; Tacrolimus; renal transplantation; immunosuppression; prevention of acute rejection
MeSH Terms: interventions — Alemtuzumab; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Campath-1H 20 mg (Experimental): Day 0: Immediately post transplant surgery patients will receive methylprednisolone 250 mg IV followed one hour later by Campath-1H 20 mg IV infusion over 3-6 hours.
  Day 1: Same protocol of Campath-1H and methylprednisolone as on Day 0.
  Day 2: No treatment
  Day 3: Initial dose of Tacrolimus 0,1 mg/kg/d (0,05 mg/kg/bid)
  till Month 6: Aim at blood level of 8-12 ng/ml (try to prevent the Tacrolimus trough level falling below 10 ng/ml in the first 3 months).
  Month 7-12: Maintain the Tacrolimus blood level at 5-8 ng/ml after 6 months.
  Interventions: Drug: Alemtuzumab
- Tacrolimus (Active Comparator): Day 0: Immediately post transplant surgery patients will receive methylprednisolone 250 mg IV followed one hour later by Campath-1H 30 mg IV infusion over 3-6 hours.
  Day 1: No treatment
  Day 2: Initial dose Tacrolimus 0.1 mg/kg/d (0.05 mg/kg.bid).
  till Month 6: Aim at blood level of 8-12 ng/ml (try to prevent the Tacrolimus trough level falling below 10 ng/ml in the first 3 months).
  Month 7-12: Maintain the Tacrolimus blood level at 5-8 ng/ml after 6 months.
  Interventions: Drug: Tacrolimus
- Campath-1H 30 mg (Experimental): Day 0: Immediately post transplant surgery patients will receive methylprednisolone 250 mg IV followed one hour later by Campath-1H 30 mg IV infusion over 3-6 hours.
  Day 1: No treatment.
  Day 2: Initial dose Tacrolimus 0.1 mg/kg/d (0.05 mg/kg.bid).
  till Month 6: Aim at blood level of 8-12 ng/ml (try to prevent the Tacrolimus trough level falling below 10 ng/ml in the first 3 months).
  Month 7-12: Maintain the Tacrolimus blood level at 5-8 ng/ml after 6 months.
  Interventions: Drug: Alemtuzumab

INTERVENTIONS:
Drug: Alemtuzumab — Day 0: Campath-1H 20 mg IV infusion over 3-6 hours
  Day 1: Campath-1H 20 mg IV infusion over 3-6 hours
  Other Names: MABCAMPATH
  Arms: Campath-1H 20 mg
Drug: Tacrolimus — Day 0: Tacrolimus will be given pre-operatively or immediately post transplant surgery. The recommended initial daily starting dose is 0,1 mg/kg/d orally (0,05 mg/kg/bid) to aim at a whole blood level of 8-12 ng/ml.
  till Month 6: Aim at blood level of 8-12 ng/ml (try to prevent the Tacrolimus trough level falling below 10 ng/ml in the first 3 months).
  Month 7-12: Maintain the Tacrolimus blood level at 5-8 ng/ml after 6 months.
  Other Names: Prograf; Advagraf
  Arms: Tacrolimus
Drug: Alemtuzumab — Day 0: Campath-1H 30 mg IV infusion over 3-6 hours
  Day 1: Campath-1H 30 mg IV infusion over 3-6 hours
  Other Names: MABCAMPATH
  Arms: Campath-1H 30 mg

SUMMARY:
The purpose of this study is to determine whether Campath following Tacrolimus monotherapy is more effective in the prevention of renal graft rejection (considering an acute rejection rate of 5% for Campath-1H/Tacrolimus and of 22% for Tacrolimus/MMF/Steroids).

DETAILED DESCRIPTION:
Major advances in immunosuppressive therapy have resulted in long-term graft survival by the use of various drug combinations.However, these combinations carry the risk of e.g. infection, malignancy, renal damage, hypertension, diabetes, hyperlipidemia, hirsutism, cushingoid facial appearance and bone necrosis.Therefore one of the major goals should be to reduce immunosuppression without increasing risk of rejections.

Based on good results of a pilot study (not a single acute rejection episode during the 18-20 months observation period despite low level of Tacrolimus and absence of steroids) this randomised trial was designed to further evaluate the safety and efficacy of Campath-1H.

ELIGIBILITY:
Inclusion Criteria:

* age 18-65
* endstage renal failure with no previous renal transplantation
* cadaveric donor
* written informed consent

Exclusion Criteria:

* pregnant or nursing women
* multi-organ transplant recipients
* live donor recipients
* re-transplants
* panel reactive antibodies (PRA) > 25%
* previous treatment with Campath-1H
* use of other investigational agents within 6 weeks
* active systemic infection
* HIV positive patient or donor
* positive lymphocyte cytotoxicity cross-match between recipient serum and donor cells
* past history of anaphylaxis following exposure to humanized monoclonal antibodies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2004-01; Primary Completion 2008-08 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Biopsy proven acute rejection episodes 6 months after transplantation (Banff Classification) | Month 6

SECONDARY OUTCOMES:
Biopsy proven acute rejection episodes 12 months after transplantation (Banff Classification) | Year 1
Time to 1st biopsy proven acute rejection episode (Banff Cl.) | Year 1
Patient and graft survival | Year 1
Number of patients who will get antilymphocyte preparation for treatment of steroid resistant acute rejection episodes | Year 1
Treatment failure defined as change from immunosuppressive protocol because of biopsy proven intractable rejection | Year 1
Adverse events (e.g. infections, PTLD) | Year 1
Creatinine clearance | Year 1

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Margreiter, Prof. Dr., Principal Investigator — Medical University for Surgery and Transplantation, Innsbruck
Locations (1):
- University Hospital Innsbruck, Innsbruck, Tyrol, Austria

REFERENCES:
- [Background] Calne R, Moffatt SD, Friend PJ, Jamieson NV, Bradley JA, Hale G, Firth J, Bradley J, Smith KG, Waldmann H. Campath IH allows low-dose cyclosporine monotherapy in 31 cadaveric renal allograft recipients. Transplantation. 1999 Nov 27;68(10):1613-6. doi: 10.1097/00007890-199911270-00032. PMID 10589966
- [Derived] Margreiter R, Klempnauer J, Neuhaus P, Muehlbacher F, Boesmueller C, Calne RY. Alemtuzumab (Campath-1H) and tacrolimus monotherapy after renal transplantation: results of a prospective randomized trial. Am J Transplant. 2008 Jul;8(7):1480-5. doi: 10.1111/j.1600-6143.2008.02273.x. PMID 18510632